CLINICAL TRIAL: NCT00119795
Title: Cooperative Lifestyle Intervention Program (CLIP)
Brief Title: Exercise and Weight Loss for Improving Mobility in Older Adults Who Are Obese
Acronym: CLIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 197; R01HL076441 (NIH); R01HL076441-01 (NIH)
Record Dates: First submitted 2005-07-06; First posted 2005-07-14 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Metabolic Syndrome X; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Metabolic Syndrome; Obesity | interventions — Exercise; Diet Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Health education control (Active Comparator): This is an education program for older adults entitles, successful aging.
  Interventions: Behavioral: Health Education Control
- Exercise Only (Experimental): Structured exercise 150 min/wk
  Interventions: Behavioral: Exercise
- Weight Loss (Experimental): Behavioral weight loss; goal of 7%
  Interventions: Behavioral: Weight Loss

INTERVENTIONS:
Behavioral: Exercise — Increase Physical Activity to 150 min/wk
  Other Names: Physical activity
  Arms: Exercise Only
Behavioral: Weight Loss — Lose 7-10% of body weight and increase physical activity to 150 min/wk
  Other Names: Diet modification
  Arms: Weight Loss
Behavioral: Health Education Control — Lectures on information relevant to successful aging
  Other Names: Attention control
  Arms: Health education control

SUMMARY:
To test the effects of exercise and weight loss on mobility disability of older overweight/obese men and women who have evidence of cardiovascular disease or the metabolic syndrome.

DETAILED DESCRIPTION:
BACKGROUND:

Older adults make up the fastest growing segment of our population. It is estimated that by the year 2030, elderly people will make up 22% of the United States population. A large portion of older adults suffers from one or more chronic conditions that could be improved by regular physical activity. Therefore, research in this age group is needed.

DESIGN NARRATIVE:

The Cooperative Lifestyle Intervention Program (CLIP) will test the effects of a physical activity intervention and a weight loss intervention on mobility disability of overweight or obese men and women who have evidence of cardiovascular disease or the metabolic syndrome. The public health relevance of the trial lies in the fact that the interventions will be delivered in conjunction with four Cooperative Extension Centers in counties surrounding Winston-Salem, North Carolina. CLIP will be designed as a three arm, randomized, controlled trial. The three 18-month treatments will include: (1) a basic health education-based control condition, (2) a group treatment program for physical activity, and (3) a lifestyle intervention designed to reduce sedentary behavior and promote weight loss. The primary aim will be to compare the effects of the three treatment arms on the change in performance on a 400-meter walk test over the course of 18 months. Secondary aims will include changes in cardiovascular risk factors, adiposity, cardiovascular fitness, physical activity, and health-related quality of life. Analyses will also be conducted to determine whether changes in the primary outcome are mediated by changes in constructs from social cognitive theory.

ELIGIBILITY:
Inclusion Criteria:

* Currently living in one of the counties surrounding Winston-Salem, NC
* Sedentary (engages in fewer than 30 minutes of moderate structured physical activity for at least 10 minutes at a time each week)
* Overweight or obese, as defined by a body mass index (BMI) greater than 25
* Fasting glucose level less than 140
* Documented evidence of an MI, PCTA, chronic stable angina, or cardiovascular surgery (coronary artery or valvular heart disease) within the 6 months prior to study entry or an ATP III diagnosis of the metabolic syndrome
* Disability defined as self-reported difficulty with walking ¼ mile, climbing stairs, lifting and carrying groceries, or performing other household chores such as cleaning and yard work
* Does not plan to move out of the county of residence for the duration of the study

Exclusion Criteria:

* Diagnosis of bipolar depression or schizophrenia (defined as self-reported treatment for these conditions)
* Currently receiving lithium or neuroleptics
* Evidence of unstable angina, symptomatic congestive heart failure, or exercise-induced complex ventricular arrhythmias
* Resting blood pressure greater than 160/100 mmHg
* Diagnosis of any of the following: Parkinson's disease; chronic liver disease (cirrhosis, chronic hepatitis, etc.); systemic rheumatic condition (rheumatoid arthritis, psoriatic arthritis, Reiter's disease, systemic lupus erythematosus, etc.); end stage renal disease; or other systemic diseases or abnormal laboratory values which would preclude participants from safely participating in the protocol or impair their ability to complete the study
* Actively being treated for cancer (other than non-melanotic skin cancer)
* Significant visual or hearing impairment that cannot be corrected and results in the inability to use the telephone or hear normal conversation
* Currently participating in or planning to participate in another medical intervention study
* Current alcohol abuse disorder or consumes more than 21 alcoholic drinks per week
* Unable to walk without assistance
* Unable to speak or read English
* Judged by the clinic staff to be unsuitable for the trial for any reason

Ages: 60 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2005-08; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
400 meter walk | Measured at 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Walter Rejeski, Principal Investigator — Wake Forest University
Locations (3):
- United States (3):
  - Guilford County, North Carolina Cooperative Extension Center, Greensboro, North Carolina
  - Davidson County Coopertive Extension, Lexington, North Carolina
  - Forsyth County Cooperative Extension Center, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brawley L, Rejeski WJ, Gaukstern JE, Ambrosius WT. Social cognitive changes following weight loss and physical activity interventions in obese, older adults in poor cardiovascular health. Ann Behav Med. 2012 Dec;44(3):353-64. doi: 10.1007/s12160-012-9390-5. PMID 22773225
- [Derived] Rejeski WJ, Brubaker PH, Goff DC Jr, Bearon LB, McClelland JW, Perri MG, Ambrosius WT. Translating weight loss and physical activity programs into the community to preserve mobility in older, obese adults in poor cardiovascular health. Arch Intern Med. 2011 May 23;171(10):880-6. doi: 10.1001/archinternmed.2010.522. Epub 2011 Jan 24. PMID 21263080